CLINICAL TRIAL: NCT07179484
Title: An Open-label, Single-arm, Multicenter Phase Ib Clinical Trial Evaluating the Efficacy, Safety, and Cellular Metabolism Kinetics of CT041 Autologous CAR-T Cell Injection as a Sequential Therapy Following First-line Treatment for Advanced Gastric/Gastroesophageal Junction Adenocarcinoma.
Brief Title: To Evaluate the Efficacy of CT041 in Sequential Treatment After First-line Treatment of Advanced Gastric/Esophagogastric Junction Adenocarcinoma
Status: Recruiting | Type: Observational
Sponsor: Beijing GoBroad Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CT041-CG4011
Record Dates: First submitted 2025-08-28; First posted 2025-09-17 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Gastroesophageal Junction Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: CT041 autologous CAR T-cell injection — The planned dose of CT041 is 2.5×108 cells. The participants are recommended to receive only a single infusion or multiple infusions (up to 3 infusions) according to the safety and efficacy data of the participants per the investigator. The dose and method of re-infusion are the same as the first infusion. Lymphodepletion pretreatment should be given before re-infusion, and the requirements before lymphodepletion pretreatment and cell infusion should also be met before re-lymphodepletion pretreatment or re-infusion.

SUMMARY:
To evaluate the efficacy of CT041 in sequential treatment after first-line treatment of advanced gastric/esophagogastric junction adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet all of the following criteria to be eligible for participation in this trial:

1. Voluntarily participate in this trial; Fully understand and be informed of this trial and sign the informed consent form; Willing to follow and able to complete all trial procedures;
2. Age 18-75 years (inclusive), male or female;
3. Pathologically confirmed unresectable locally advanced or metastatic advanced gastric/esophagogastric junction (G/GEJ) adenocarcinoma;
4. Immunohistochemical (IHC) staining of tumor tissue sample is CLDN18.2 positive, defined as staining intensity ≥ 2 + in at least 40% of tumor cells;
5. Completed 12 weeks of first-line therapy according to clinical guidance, without disease progression as assessed by the investigator:

   Permitted treatment regimens include: fluoropyrimidine + platinum (± taxane) regimen chemotherapy, with or without immunotherapy or zolbetuximab. Other treatment regimens may be allowed to be included after discussion between the investigator and medical monitor of the collaborator; For the treatment regimen of every 2 weeks, 6 cycles should be completed, and for the treatment regimen of every 3 weeks, 4 cycles should be completed; According to the investigator's assessment and decision, participants without disease progression after at least 6 weeks of first-line treatment can undergo apheresis after meeting other eligibility criteria;
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (within 7 days prior to apheresis);
7. Adequate venous access for apheresis and no other contraindications for apheresis.
8. Laboratory test results within 7 days prior to apheresis should meet the following criteria (a repeat test within one week is allowed, if still not meeting the criteria, it will be considered a screening failure):

   1. Blood routine (without transfusion, platelet transfusion, colony-stimulating factor, platelet growth factor and other supportive treatment within 7 days before test, except recombinant human erythropoietin): absolute neutrophil count (ANC) ≥ 1.5×109/L, lymphocyte (LY) ≥ 0.5×109/L, platelet (PLT) ≥ 75×109/L, hemoglobin (Hb) ≥ 9.0 g/dL. The results of blood routine test within 24 hours before apheresis should also meet the above criteria.
   2. Blood chemistry: endogenous creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula), alanine aminotransferase (ALT) ≤ 2.5×upper limit of normal (ULN), aspartate aminotransferase (AST) ≤ 2.5×ULN, total bilirubin ≤ 2×ULN; serum amylase ≤ 2.0×ULN; alkaline phosphatase ≤ 2.5×ULN; AST, ALT and alkaline phosphatase ≤ 5 × ULN if there is bone metastasis or liver metastasis;
   3. Prothrombin time (PT) prolongation ≤ 4 seconds.
9. Female participants of childbearing potential (WOCBP) must have a negative serum pregnancy test at screening and be willing to use highly effective and reliable contraception (< 1% failure rate per year) for at least 12 months after receiving trial treatment and egg donation is absolutely prohibited during this period.
10. Male participants who are sexually active with a female of childbearing potential, who have not had a vasectomy, must agree to practice abstinence or use highly effective and reliable contraception (failure rate < 1% per year) for at least 12 months after receiving trial treatment and sperm donation is prohibited during this period.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from this trial:

1. Presence of a known tumor tissue with high HER2 expression;
2. Presence of gastrointestinal bleeding/perforation/obstruction or significant risk with these, including but not limited to anastomotic recurrence involving the full thickness of gastric wall, deep large ulcer, unstable/active ulcer, history of gastrointestinal bleeding/perforation/obstruction within 3 months (excluding those with surgical resection of the lesion leading to such event);
3. Participants who have previously received any anti-tumor therapy other than the first-line treatment regimen for G/GEJ adenocarcinoma allowed in this trial (see Item 5 of the inclusion criteria), including any other systemic anti-tumor drugs, any radiotherapy or interventional therapy, etc.;
4. Systemic anti-tumor treatment for G/GEJ adenocarcinoma within 21 days (or within 5 half-lives of the drug, whichever is shorter) prior to apheresis;
5. Major surgery (excluding cataract surgery and other surgery requiring local anesthesia) or significant traumatic injury within 4 weeks prior to apheresis and has not adequately recovered from toxicity and/or complications;
6. Previously received any genetic engineering modified cell therapy (such as CAR-T cells, TCR-T cells, etc.);
7. Toxicities from previous treatment that have not recovered to Common Terminology Criteria for Adverse Events (CTCAE) v5.0 ≤ Grade 1, excluding alopecia, pigmentation, peripheral neuropathy, other events that, at the discretion of the investigator, do not affect the tolerability of the participant to the trial intervention, and laboratory abnormalities allowed in this trial.

   Note: Participants with non-clinically significant Grade 2 AE may be allowed to be included in the trial after discussion with medical monitor of the collaborator;
8. Positive serology for human immunodeficiency virus (HIV), Treponema pallidum, or hepatitis C virus (HCV). Participants with positive HCV antibody but negative HCV RNA can be enrolled;
9. Any active infection, including but not limited to active tuberculosis infection, active HBV infection (including hepatitis B surface antigen [HBsAg] positive, or hepatitis B core antibody [HBcAb] positive with HBV DNA above the lower limit of the trial center lab), and infection with other pathogens requiring systemic treatment. Participants receiving prophylactic anti-infective therapy may be enrolled at the discretion of the investigator;
10. Participants with clinically significant thyroid dysfunction or severe complications that are not suitable for participation in this trial at the discretion of the investigator. Participants with stable thyroid function after treatment can be considered for enrollment;
11. Received systemic corticosteroids within 14 days prior to apheresis. Recent or current use of inhaled or topical skin corticosteroids and physiologic dose replacement therapy may be enrolled;
12. Need for long-term anticoagulation/antiplatelet therapy (e.g. Warfarin, heparin, rivaroxaban, aspirin, dipyridamole, clopidogrel, etc.). Participants receiving prophylactic anticoagulation to maintain patency of venous access devices may be enrolled;
13. Allergy to fludarabine, cyclophosphamide, nab-paclitaxel, tocilizumab and other related drugs, or known allergy to components of CT041 cell infusion preparation (such as albumin or dimethyl sulfoxide [DMSO], etc.), or history of severe allergy in the past;
14. Presence of known or suspected central nervous system metastases;
15. Presence of central type or extensive lung metastasis, or extensive liver metastasis, or extensive bone metastasis;
16. Abdominal/pleural effusion with clinical symptoms or requiring special treatment, such as repeated drainage, abdominal/pleural drug perfusion, etc. (participants with small amount of ascites/pleural effusion that can be detected by imaging examination can be considered for enrollment);
17. Participants who have previously received organ transplantation or allogeneic hematopoietic stem cell transplantation, or are awaiting organ transplantation;
18. Vaccination with live or live attenuated vaccines within 4 weeks prior to apheresis or planned during the trial;
19. Presence of active autoimmune diseases, including but not limited to rheumatoid arthritis, systemic lupus erythematosus, autoimmune hepatitis, interstitial lung disease, inflammatory bowel disease, antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, multiple sclerosis, glomerulonephritis, etc.; And currently receiving or requiring long-term immunosuppressant therapy during the trial;
20. Presence of any of the following cardiovascular diseases: uncontrolled congestive heart failure (New York Heart Association [NYHA] Class III-IV), cardiac dysfunction [left ventricular ejection fraction (LVEF) < 50%], myocardial infarction within the last 6 months, poorly controlled arrhythmia, unstable angina, poorly controlled hypertension (blood pressure > 160 mmHg/100 mmHg), hypotension that is symptomatic or requires vasopressor medication, and other diseases or test abnormalities that are deemed inappropriate for participation in the trial by the investigator. Discussion with medical monitor of the collaborator is recommended if necessary;
21. Pulmonary diseases that are not suitable for participation in this trial as assessed by the investigator, including but not limited to: chronic obstructive pulmonary disease, pulmonary embolism, interstitial lung disease, clinically significant abnormal pulmonary function test, etc. Discussion with medical monitor of the collaborator is recommended if necessary;
22. Oxygen saturation (SaO2) ≤ 95% without oxygen inhalation (finger oxygen detection method is accepted);
23. Presence of clinically significant neurological disorders, psychiatric disorders or abnormal neurological examination results;
24. As assessed by the investigator, the participant has poor glycemic control under adequate treatment or has experienced relevant complications;
25. Presence of any clinicopathological features, other diseases, metabolic disorders, signs or abnormal examination results that prohibit the trial intervention, affect the interpretation of the results, preclude CT041 infusion, or are at high risk of serious complications after infusion, and are assessed as unsuitable for participation by the investigator;
26. Uncured malignant tumor other than G/GEJ cancer in the past 5 years or at the same time; Except for adequately treated basal cell carcinoma of the skin, carcinoma in situ of the cervix and other malignancies with very low risk of metastasis or death;
27. Pregnant or lactating females;
28. Participants who are unable or unwilling to comply with the requirements of the clinical trial protocol as assessed by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with unresectable locally advanced or metastatic gastric/esophagogastric junction adenocarcinoma who have not progressed after 12 weeks of first-line therapy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-10-22 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of CT041 in sequential treatment after first-line treatment of advanced gastric/esophagogastric junction adenocarcinoma | For 18 months
  Progression-free survival (PFS)
peak CAR copy number (Cmax) | 12 months
  peak CAR copy number (Cmax)

SECONDARY OUTCOMES:
Event-free survival (EFS) | Approximately 24 months
  Event-free survival (EFS)
Overall survival (OS) | Approximately 24 months
  Overall survival (OS)
Incidence, type, and severity of adverse events | Signing ICF to CT041 infusion 15 years later
  Incidence, type and severity of adverse events, including:
  Adverse events (AEs); Adverse events of special interest (AESIs); Serious Adverse Events (SAEs), etc.
Objective Response Rate（ORR） | Approximately 24 months
  Objective Response Rate（ORR）
Disease control rate（DCR） | Approximately 24 months
  Disease control rate（DCR）
Duration of response (DOR) | Approximately 24 months
  Duration of response (DOR)
Duration of disease control (DDC) | Approximately 24 months
  Duration of disease control (DDC)
Progression-free survival-1 (PFS-1) | Approximately 24 months
  Progression-free survival-1 (PFS-1)
Overall survival-1 (OS-1) | Approximately 24 months
  Overall survival-1 (OS-1)
CAR copy number, time to peak CAR copy number (Tmax) | Approximately 12 months
  CAR copy number, time to peak CAR copy number (Tmax)
area under the curve (AUC) and cell persistence (Tlast) after CT041 infusion | Approximately 12 months
  area under the curve (AUC) and cell persistence (Tlast) after CT041 infusion

CONTACTS AND LOCATIONS:
Locations (1):
- BeijingGoBroadH, Beijing, China

IPD SHARING:
Plan to Share IPD: No